CLINICAL TRIAL: NCT04386265
Title: The Compassionate Use of Hyperbaric Oxygen Therapy in the Treatment of COVID-19
Brief Title: Compassionate Use of Hyperbaric Oxygen Therapy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: SerenaGroup Research Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: HBOT-COVID-19
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
Keywords: COVID-19; Mechanical Ventilation; Hyperbaric Oxygen Therapy; Patient Registry
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational patient registry of COVID-19 patients treated with HBOT.

DETAILED DESCRIPTION:
The retrospective analysis will focus on the reduction in need for mechanical ventilation in COVID-19 patients. The information will be gathered prospectively. Data will be collected from the patients' medical record, including medical notes and data recorded into the study database.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with COVID-19.
* The clinical decision to use HBOT is independent of the decision to participate in registry.
* A signed and dated informed consent form for the off-label use of Hyperbaric Oxygen Therapy specific to the institution where treatment is rendered.
* Subject is willing and able to comply with instructions and scheduled visits.

Exclusion Criteria:

* The Subject has other concurrent conditions that in the opinion of the Investigator may compromise patient safety.
* The patient has an untreated pneumothorax.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-05-11 (Estimated); Study Completion 2022-05-11 (Estimated)

PRIMARY OUTCOMES:
Gather information on patients treated with hyperbaric oxygen therapy | 24 months
  Collect information on the reduction in need for mechanical ventilation in COVID-19 patients.

SECONDARY OUTCOMES:
Gather information on adverse events | 24 months
  Follow adverse events associated with the treatment of COVID-19 related to HBOT

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Serena, MD, Study Director — SerenaGroup, Inc.
Locations (11):
- United States (10):
  - White River Wound Healing Center, Batesville, Arkansas
  - Community Hospital, Monterey, California
  - Innovative Healing Systems, Tampa, Florida
  - Decatur Memorial Hospital, Decatur, Indiana
  - Providence Medical Wound Care Center, Kansas City, Kansas
  - West Jefferson Medical Center, Marrero, Louisiana
  - The Wound Treatment Center, Opelousas, Louisiana
  - Christus Shreveport Bossier Hyperbaric & Wound Care Center, Shreveport, Louisiana
  - Ascension Providence Rochester Hospital Wound Care Center, Rochester, Michigan
  - CHI, Chattanooga, Tennessee
- Klinika Baromedical, Poznan, Greater Poland Voivodeship, Poland